CLINICAL TRIAL: NCT06537440
Title: Electroacupuncture for the Management of Opioid-Induced Constipation in Patients With Cancer: a Study Protocol for a Single-Center, Single-Blind, Randomized Controlled Trial
Brief Title: Electroacupuncture for Opioid-Induced Constipation in Cancer Patients: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Kong Fanming, chairman of section, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TYLL2023[Z]字012
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Constipation, Opioid-Induced; Cancer
Keywords: Opioid-related constipation; cancer; electroacupuncture; sham electroacupuncture control
MeSH Terms: conditions — Opioid-Induced Constipation; Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Due to the specific nature of acupuncture clinical research, it is difficult to accomplish double blinding of subjects and operators, so this trial was blinded to subjects, outcome assessors, and statisticians only. To assess the success of blinding, all patients who received acupuncture were asked to guess their group allocation five minutes after the completion of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental): In the EA group, acupoints TE6, ST36, ST25, and CV12 will be used. With the participant lying supine, the skin will be disinfected before needle insertion. For ST25 and CV12, 0.25×50 mm needles will be inserted vertically into the abdominal muscle layer until Deqi is achieved. For TE6 and ST36, needles measuring 0.25 × 40 mm and 0.25 × 50 mm, respectively, will be inserted vertically to depths of approximately 15 mm and 35 mm. Manual stimulation will be applied using three uniform lifting, thrusting, and twirling manipulations to elicit Deqi. Electrodes from an SDZ-V EA device will then be attached to TE6 and ST36. A continuous 20 Hz electrical stimulation at 0.5-4 mA (based on tolerance) will be applied for 30 minutes.
  Interventions: Other: Electroacupuncture
- Sham Acupuncture group (Sham Comparator): Participants in the SA group will receive shallow needle insertion (2-3 mm) at non-acupoint sites near TE6, ST36, ST25, and CV12. After skin disinfection, 0.25×40 mm sterile needles will be inserted without manual stimulation or eliciting Deqi. The sham electrode wires attached to the pseudo-TE6 and ST36 points will appear identical to those used in the EA group; however, the internal metal conductors will be cut to prevent current transmission. As a result, although the electrical stimulation device will display an active status (with indicator lights on and sound output), no actual electrical current will be delivered. The stimulation parameters and treatment duration will mirror those used in the EA group.
  Interventions: Other: Electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture — Electroacupuncture TE6 Zhigou (double), ST36 Zusanli (double), ST25 Tianshu (double), CV12 Zhongwan

SUMMARY:
The primary objective of this trial is to evaluate the efficacy and safety of electroacupuncture in the management of opioid-induced constipation in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of OIC based on the Rome IV Criteria: Participants must meet the following criteria for OIC: Constipation or worsening of constipation symptoms during opioid use or dose changes, with at least two of the following symptoms: 1. at least 25% of bowel movements are labored; 2. at least 25% of bowel movements are dry ball or hard stools; 3. at least 25% of bowel movements are incomplete; 4. at least 25% of bowel movements have anal rectal obstruction and/or blockage in at least 25% of the bowel movements; 5. at least 25% of the bowel movements required manual assistance (e.g., finger-assisted defecation, pelvic floor support); 6. less than 3 bowel movements per week; (2) the rare occurrence of loose stools when laxatives were not used.
2. Rare occurrence of loose stools without the use of laxatives;
3. History of OIC symptoms for at least 1 week prior to enrollment;
4. Age: Participants must be aged between 18 and 85 years;
5. Cancer Status: Participants must have stable cancer with a life expectancy of greater than 6 months;
6. ECOG Performance Status: Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3;
7. Stable Opioid Maintenance: Participants must have been receiving a relatively stable opioid regimen for at least 2 weeks prior to screening, with a daily morphine equivalent dose (MED) ranging from 30 mg to 1000 mg. Additionally, opioid treatment is expected to continue for at least 10 weeks;
8. Bowel Movement Frequency: In the absence of laxative use, participants must have fewer than two spontaneous bowel movements (SBMs) per week;
9. Ability to Take Oral Medications: Participants must be capable of swallowing oral medications, food, and beverages;
10. Informed Consent: Participants must voluntarily consent to participate in the trial and provide signed informed consent;
11. Exclusion of Gastrointestinal Motility Agents: Participants must not have used any gastrointestinal motility-promoting drugs within 1 week prior to randomization.

Exclusion Criteria:

1. Significant Bowel Dysfunction due to Gastrointestinal or Other Structural Abnormalities: Participants diagnosed with clinically significant bowel dysfunction resulting from gastrointestinal or related structural abnormalities (excluding OIC), such as inflammatory bowel disease, rectal prolapse, gastrointestinal obstruction, peritoneal metastases, or peritoneal tumors;
2. Recent History of Abdominal Surgery: Participants with a history of gastrointestinal or abdominal surgery, or abdominal adhesions within 1 month prior to screening; or a history of bowel obstruction within 3 months prior to screening;
3. Active Gastrointestinal Conditions: Diagnosis of active diverticular disease, severe hemorrhoids, anal fissures, or artificial rectum or anus;
4. Presence of Abdominal Catheters or Feeding Tubes: Participants with abdominal catheters or feeding tubes in place;
5. Pelvic Diseases Affecting Bowel Transit: Participants diagnosed with pelvic diseases known to significantly affect bowel transit (e.g., ≥2nd degree uterine prolapse, uterine fibroids ≥5 cm located in the posterior uterus);
6. Recent or Planned Chemotherapy: Participants who received a new chemotherapy regimen within 14 days of screening, or who plan to receive such treatment during the study period;
7. Recent or Planned Radiotherapy: Participants who received radiotherapy within 28 days prior to screening, or who plan to undergo radiotherapy during the study period;
8. Recent Gastrointestinal Surgery or Interventions: Participants who have undergone or are scheduled to undergo surgeries or interventions within 28 days of screening that could significantly affect gastrointestinal function or are expected to prevent completion of the trial;
9. Uncontrolled Medical Conditions: Participants with uncontrolled hyperthyroidism, severe hypertension, cardiovascular disease, systemic infections, or coagulation disorders (e.g., hypercoagulability or bleeding tendencies);
10. Excessive Use of Opioids Due to Acute Pain: Participants who have required more than four additional doses of opioid analgesics per day for more than 3 consecutive days during the baseline period due to acute pain, or those who have modified their opioid maintenance regimen during this period;
11. Severe Cancer Pain Unresponsive to Opioids: Participants who experience severe cancer-related pain despite standard opioid therapy (e.g., average daily pain intensity of 7-10 on the Numerical Rating Scale [NRS], where 0 is "no pain" and 10 is "the worst pain possible");
12. History of Opioid Discontinuation Due to Severe Adverse Events: Participants with a history of opioid discontinuation due to severe adverse events, or those expected to discontinue opioid use due to potential risks of adverse events;
13. Recent Use of Opioid Antagonists: Participants who have received opioid receptor antagonists within 1 month prior to screening;
14. Inability to Provide Informed Consent: Participants who are unconscious, psychotic, or unable to express subjective symptoms. (As acupuncture is an invasive procedure requiring 30 minutes per session, such participants will be excluded for safety reasons.);
15. Bleeding Disorders: Participants with bleeding disorders, as acupuncture involves skin penetration, and individuals with bleeding tendencies are at increased risk of complications;
16. Recent Acupuncture Treatment: Participants who have received acupuncture treatment within 3 months prior to screening;
17. Participation in Other Clinical Trials: Participants who have participated in or are currently participating in another clinical trial within the past 3 months;
18. Other Medical or Treatment Conditions: Any other participants deemed by the investigator to be unsuitable for the study due to concomitant treatments or medical findings.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
The proportion of responders. | At the end of the 1-week treatment period
  Patients will have at least three spontaneous bowel movements (SBMs) per week during the treatment period and an increase of at least one SBM from baseline during the treatment period. A bowel movement can only be described as SBM if it has occurred without any intervention to assist in defecation in the past 24 hours.

SECONDARY OUTCOMES:
The weekly mean number of SBMs | (1)Assessments will be conducted at baseline, Week 1 (end of treatment), Week 2, and Week 3 (follow-up).
Weekly mean CSBMs | Assessments will be conducted at baseline, Week 1 (end of treatment), Week 2, and Week 3 (follow-up).
  CSBMs are defined as SBMs accompanied by a self-reported sense of complete evacuation
Weekly mean Bristol Stool Form Scale (BSFS) score | Assessments will be conducted at baseline, Week 1 (end of treatment), Week 2, and Week 3 (follow-up).
  Stool consistency will be assessed using the Bristol Stool Form Scale (BSFS), a validated 7-point scale ranging from Type 1 (hard, lumpy) to Type 7 (watery). Types 3-5 are considered normal
Weekly mean straining of constipation scores | Participants will complete daily scores; weekly mean scores will be will be calculated at baseline, Week 1 (end of treatment), Week 2, and Week 3 (follow-up).
  Straining will be self-rated using a 5-point scale: 0 = not at all difficult, 1 = a little bit, 2 = moderately, 3 = quite a bit, and 4 = extremely difficult.
Use of Rescue Medications or Other Bowel Support Measures. | The proportion of participants requiring rescue interventions (e.g., laxatives, enemas, suppositories) and the mean frequency of use per week will be recorded from the start of treatment (Day 0) through the end of follow-up (Day 21).
The Patient Assessment of Constipation-Symptom (PAC-SYM) scores | The validated Chinese version of PAC-SYM will be used, assessed at baseline, Week 1, and Week 3.
  Changes in symptom severity will be assessed using the Patient Assessment of Constipation-Symptom (PAC-SYM) questionnaire, a 12-item instrument evaluating symptoms over the past 2 weeks. It includes abdominal (4 items), rectal (3 items), and stool (5 items) subscales. Each item is scored from 0 (no symptom) to 4 (very severe), with lower scores indicating milder symptoms. Subscale and total scores are calculated as the mean of completed items.
The Patient Assessment of Constipation-Quality of Life (PAC-QOL) scores | The validated Chinese version will be administered at baseline, Week 1, and Week 3.
  The Patient Assessment of Constipation-Quality of Life (PAC-QOL) questionnaire assesses the impact of constipation on daily functioning and well-being over the past 2 weeks. It contains 28 items across four subscales: physical discomfort (items 1-4), psychosocial discomfort (items 5-12), worries/concerns (items 13-23), and satisfaction (items 24-28). Each item is scored from 0 (not at all) to 4 (extremely), with lower scores indicating better quality of life.
Patients' global assessment of treatment efficacy. | Assessment will be conducted on Day 7.
  Participants will rate their perceived treatment efficacy using a 7-point global assessment scale: 1 = markedly worse, 2 = moderately worse, 3 = slightly worse, 4 = no change, 5 = slightly improved, 6 = moderately improved, 7 = markedly improved. This scale has demonstrated reliability and ease of use.
The changes in gut microbiota and microbial metabolites. | Fecal samples were collected at baseline and after the 1-week treatment.
  16S ribosomal RNA (16S rRNA) gene sequencing was performed to evaluate the composition, diversity, and relative abundance of gut microbial communities.In parallel, untargeted metabolomic profiling using liquid chromatography-mass spectrometry (LC-MS) will be conducted to identify and quantify microbial metabolites.

CONTACTS AND LOCATIONS:
Locations (1):
- First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided